CLINICAL TRIAL: NCT00128622
Title: A Phase I Study of Regulatory T Cell Depletion With Denileukin Diftitox Followed by Active Immunotherapy With Autologous Dendritic Cells Infected With CEA-6D Expressing Fowlpox-Tricom in Patients With Advanced or Metastatic Malignancies Expressing CEA
Brief Title: Denileukin Diftitox Followed by Vaccine Therapy in Treating Patients With Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Kim Lyerly (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, H. Kim Lyerly, Professor, Gen & Thor Surgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000437795; DUMC-NCI-7042; NCI-7042
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Breast Cancer; Colorectal Cancer; Lung Cancer; Pancreatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: male breast cancer; recurrent breast cancer; stage IV breast cancer; recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer; recurrent pancreatic cancer; extensive stage small cell lung cancer; recurrent non-small cell lung cancer; recurrent small cell lung cancer; stage IV non-small cell lung cancer; unspecified adult solid tumor, protocol specific; stage IV pancreatic cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Breast Neoplasms, Male; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — denileukin diftitox

ARMS (1):
- Denileukin Diftitox plus vaccine (Experimental): This is a single arm Phase I safety study.
  Interventions: Biological: denileukin diftitox; Biological: recombinant fowlpox-CEA(6D)/TRICOM vaccine; Biological: therapeutic autologous dendritic cells

INTERVENTIONS:
Biological: denileukin diftitox
Biological: recombinant fowlpox-CEA(6D)/TRICOM vaccine
Biological: therapeutic autologous dendritic cells

SUMMARY:
RATIONALE: Combinations of biological substances in denileukin diftitox may be able to carry cancer-killing substances directly to the cancer cells. Vaccines made from a gene-modified virus and a person's white blood cells may help the body build an effective immune response to kill cancer cells. Giving denileukin diftitox together with vaccine therapy may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects of giving denileukin diftitox together with vaccine therapy in treating patients with metastatic cancer that expresses carcinoembryonic antigen.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and feasibility of two different schedules of denileukin diftitox followed by active immunotherapy comprising autologous dendritic cells infected with recombinant fowlpox-CEA(6D)-TRICOM vaccine in patients with metastatic CEA-expressing malignancies.

Secondary

* Determine the immune response to this regimen in these patients.
* Determine, preliminarily, clinical response rate and/or time to progression in patients with assessable disease treated with this regimen.

OUTLINE: Patients undergo leukapheresis for collection of peripheral blood mononuclear cells (PBMCs). PBMCs are cultured with sargramostim (GM-CSF) and interleukin-4 for the production of dendritic cells( DC). DC are mixed with recombinant fowlpox-TRICOM to produce the vaccine. Patients are assigned to 1 of 2 cohorts according to timing of study enrollment.

* Cohort 1: Patients receive denileukin diftitox IV over at least 15 minutes once in week 0 and vaccine therapy comprising autologous DC infected with recombinant fowlpox-CEA (6D)-TRICOM vaccine intradermally and subcutaneously once in weeks 0 (beginning 4 days after the denileukin diftitox infusion), 3, 6, and 9. If < 2 of 6 patients experience dose-limiting toxicity, a second cohort of patients is enrolled.
* Cohort 2: Patients receive denileukin diftitox as in cohort 1 once in weeks 0, 3, 6, and 9 and vaccine as in cohort 1.

In both cohorts, treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed annually for up to 15 years.

PROJECTED ACCRUAL: A total of 6-12 patients (6 per cohort) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy

  * Metastatic disease
* Tumor expresses carcinoembryonic antigen (CEA), as evidenced by any of the following:

  * At least 50% of tumor expresses CEA by immunohistochemistry (IHC) with ≥ a moderate intensity of staining
  * Peripheral blood CEA level > 5.0 ng/mL
  * Tumor known to be universally CEA-positive (e.g., colon or rectal cancer)
* Measurable or evaluable disease
* Received or refused prior therapy with a possible survival or palliative benefit AND meets the following disease-specific criteria:

  * Patients with colorectal cancer must have experienced disease progression during ≥ 1 prior palliative chemotherapy regimen for metastatic disease comprising 1 of the following regimens:

    * Fluorouracil or capecitabine AND oxaliplatin
    * Fluorouracil or capecitabine AND irinotecan
    * Chemotherapy in combination with bevacizumab
  * Patients with breast cancer must have experienced disease progression during ≥ 1 prior palliative chemotherapy regimen for metastatic disease comprising 1 of the following regimens:

    * Anthracycline- or taxane-based chemotherapy
    * Chemotherapy AND trastuzumab (Herceptin®) (required for patients with tumors overexpressing HER2/neu (i.e., 3+ by IHC or positive by fluorescence in situ hybridization [FISH])
  * Patients with lung cancer must have experienced disease progression during ≥ 1 prior palliative chemotherapy regimen for metastatic disease comprising 1 of the following regimens:

    * Platinum-based (e.g., cisplatin or carboplatin) chemotherapy (for chemotherapy-naive patients only)
    * Taxane-based (e.g., docetaxel or paclitaxel) chemotherapy OR vinorelbine (for patients who received prior chemotherapy)
  * Patients with pancreatic cancer must have experienced disease progression during prior chemotherapy, including gemcitabine
  * Patients with other malignancies must have experienced disease progression after prior first-line therapy that would confer a survival or palliative benefit, if such a therapy exists

    * Patients who experienced disease progression during prior first-line palliative chemotherapy must be advised regarding second-line therapy before study enrollment
* Previously resected brain metastases allowed provided there is no evidence of brain metastasis within the past month by MRI or CT scan
* No requirement for further systemic chemotherapy for ≥ 3 months
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* Karnofsky 70-100%

Life expectancy

* More than 6 months

Hematopoietic

* WBC ≥ 3,000/mm^3
* Hemoglobin ≥ 9 g/dL (transfusion or epoetin alfa allowed)
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin < 1.5 mg/dL (≤ 2.0 mg/dL for patients with Gilbert's syndrome)
* SGOT and SGPT < 1.5 times upper limit of normal
* Albumin ≥ 3.0 g/dL
* No active acute or chronic viral hepatitis

  * Hepatitis B surface antigen negative
  * Hepatitis C negative
* No other hepatic disease that would preclude study treatment

Renal

* Creatinine < 1.5 mg/dL
* No active acute or chronic urinary tract infection

Cardiovascular

* No New York Heart Association class III-IV cardiac disease

Immunologic

* HIV negative
* No history of autoimmune disease*, including, but not limited to, the following:

  * Inflammatory bowel disease
  * Systemic lupus erythematosus
  * Ankylosing spondylitis
  * Scleroderma
  * Multiple sclerosis
* No active cytomegalovirus (CMV) disease

  * Patients with CMV-seropositivity are eligible
* No other active acute or chronic infection
* No history of allergies to eggs or any component of the study vaccine, denileukin diftitox, or diphtheria toxin NOTE: *Patients with a positive anti-nuclear antibody (ANA) ≤ 1:256 with no other evidence of autoimmune disease are eligible

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 months after completion of study treatment
* No acute or chronic skin disorder that would preclude study treatment
* No other malignancy within the past 5 years except nonmelanoma skin cancer, controlled carcinoma in situ of the cervix, or controlled superficial bladder cancer
* No psychological or medical impediment that would preclude study compliance
* No other serious acute or chronic illness that would preclude study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* Prior vaccine, dendritic cell, or CEA-targeted immunotherapy allowed
* At least 4 weeks since prior and no other concurrent immunotherapy
* Concurrent palliative single-agent trastuzumab for breast cancer allowed provided patient has been on therapy for ≥ 3 months before study entry

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior and no concurrent chemotherapy

Endocrine therapy

* At least 4 weeks since prior hormonal therapy
* At least 6 weeks since prior steroid therapy except steroids used as premedication for chemotherapy or contrast-enhanced studies
* No concurrent steroids, including corticosteroids administered to manage toxic effects from dendritic cell or denileukin diftitox administration
* Concurrent palliative endocrine therapy for breast cancer allowed provided patient has been on therapy for ≥ 3 months before study entry

Radiotherapy

* At least 4 weeks since prior and no concurrent radiotherapy

Surgery

* See Disease Characteristics

Other

* Recovered from all prior therapy
* At least 4 weeks since prior investigational drugs or procedures
* At least 4 weeks since other prior therapy
* No other concurrent immunosuppressive therapy (e.g., azathioprine or cyclosporine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-09; Primary Completion 2007-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Safety as measured by rate of adverse events during study drug treatment | 3 months

SECONDARY OUTCOMES:
Rate of immune response as measured by ELISPot at week 10 | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Morse, MD, Study Chair — Duke Cancer Institute
Locations (2):
- United States (2):
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Duke Comprehensive Cancer Center, Durham, North Carolina

REFERENCES:
- [Background] Schonfeld K, Mahnke K, Schallenberg S, et al.: Treatment of melanoma bearing individuals with ONTAK® depletes regulatory T cells resulting in an augmented immune response following vaccination. [Abstract] J Invest Dermatol 126 (Suppl S3): A-594, s101, 2006.
- [Derived] Morse MA, Hobeika AC, Osada T, Serra D, Niedzwiecki D, Lyerly HK, Clay TM. Depletion of human regulatory T cells specifically enhances antigen-specific immune responses to cancer vaccines. Blood. 2008 Aug 1;112(3):610-8. doi: 10.1182/blood-2008-01-135319. Epub 2008 Jun 2. PMID 18519811